CLINICAL TRIAL: NCT02804880
Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2016: a Single-blind Cluster Randomized Controlled Trial on High Intensity Active Referral and Simple Text Messaging to Achieve Abstinence
Brief Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2016
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QTW2016
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-10

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Quit to Win; Brief intervention; Personalized active referral; Instant messaging; SMS; Smoking Cessation Intervention
MeSH Terms: conditions — Smoking Cessation | interventions — corticosteroid hormone-induced factor; Referral and Consultation; Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): HAR + AWARD + Referral Card + A4 leaflet
  Interventions: Behavioral: HAR; Behavioral: AWARD; Other: Referral card; Other: A4 leaflet
- Group B (Experimental): LTM + AWARD + Referral Card + A4 leaflet
  Interventions: Behavioral: LTM; Behavioral: AWARD; Other: Referral card; Other: A4 leaflet
- Group C (Active Comparator): Brief advice + 12-page booklet
  Interventions: Behavioral: Brief advice; Other: 12-page booklet

INTERVENTIONS:
Behavioral: HAR — Smokers will be introduced to various smoking cessation (SC) services in Hong Kong (using the referral card) and be motivated to use the services. Field research staff will assist on-site booking SC services for smokers. Tailored messages, including: harm of smoking, benefit of smoking cessation, importance of adherence to smoking cessation appointment and encouragement on abstinence will be sent via instant messaging (IM) services (e.g. WhatsApp, WeChat) to smokers after initial contact.
  Other Names: Higher intensity and personalized active referral (HAR)
  Arms: Group A
Behavioral: LTM — Fix-schedule SMS messages will be sent to encourage them to book the smoking cessation services appointment. Smokers are required to book the SC appointments by themselves.
  Other Names: Low-intensity text messaging on using SC services (LTM)
  Arms: Group B
Behavioral: AWARD — Ask about smoking history, Warn about the high risk of smoking, Advise to quit as soon as possible, Refer to the smoking cessation services, and Do it again: to repeat the intervention during tel. follow-ups.
  Other Names: Ask, Warn, Advise, Refer, Do-it-again
  Arms: Group A; Group B
Other: Referral card — The 3-folded "Smoking Cessation Services" card consists of brief information and highlights of existing smoking cessation services, contact methods, motivation information and strong supporting messages or slogans.
  Other Names: Smoking Cessation Service Card
  Arms: Group A; Group B
Other: A4 leaflet — The 2-side color printed A4 leaflet, which systematically covers the most important messages to motivate smoking cessation
  Other Names: Brief leaflet on health warning and smoking cessation
  Arms: Group A; Group B
Behavioral: Brief advice — Very brief, minimal and general smoking cessation advice
  Other Names: Brief smoking cessation advice
  Arms: Group C
Other: 12-page booklet — 12-page smoking cessation self-help booklet
  Other Names: 12-page smoking cessation booklet
  Arms: Group C

SUMMARY:
The present study will examine (1) the effectiveness of personalised active referral to smoking cessation (SC) services and text messaging on encouraging SC services (2) explore the use of CBPR model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

DETAILED DESCRIPTION:
Although smoking prevalence is decreasing in Hong Kong, there are still 641,300 daily smokers (10.5%; Census and Statistics Department, 2015) and half will be killed by smoking (Lam, 2012) which accounts for over 7,000 deaths per year (Lam, Ho, Hedley, Mak, & Peto, 2001). Smoking also accounts for a large amount of medical cost, long-term care and productivity loss of US$688 million (0.6% Hong Kong GDP) (Census & Statistics Department, 2001; McGhee et al., 2006) . Smoking is a highly addictive behavior and it is difficult for smokers with strong nicotine dependence to quit without assistance. On the other hand, reaching and helping the many smokers who have no intention to quit is a challenge, because they are unlikely to seek professional help from smoking cessation services.

The Quit and Win programme provides an opportunity to reach and encourage a large group of smokers to make quit attempt and maintain abstinence. The Quit and Win model posits that smokers participating in the contest will have higher motivation to quit with incentives and better social support (Cahill & Perera, 2011). Studies have found that such quitting contests or incentive programs appeared to reach a large number of smokers and demonstrated a significantly higher quit rate for the quit and win group than for the control group (Cahill & Perera, 2015).

Smoking cessation services in Hong Kong are under-used with most of the adult daily smokers (79.6%) who had never used smoking cessation services (Census and Statistics Department, 2015). Among these smokers, only 2.4% were willing to use the services. Our previous RCT in previous QTW Contest 2015 evaluated the effects of low-intensity active referral (LAR) vs. very brief general SC advice (VBA) on quitting. LAR included onsite AWARD counselling and collection of smokers' personal contact information for SC services providers to connect with the smokers. Findings at 3-month follow-up of this RCT suggested the LAR intervention resulted in significantly higher self-reported quit rate than VBA in the control group (18.7% vs 14.0%. P<0.001).

It is warranted to evaluate if a higher intensity active referral (HAR) and/or text messaging on encouraging SC services use can achieve even higher quit rate when compared with only VBA is given in the control group. Noted the use of text-messaging is the cheaper method than HAR. By using the same design of control group in QTW 2015, we can combine and compare the 2 years QTW intervention of HAR, LAR and text-messaging using network meta-analysis. This will contribute to finding out a more cost-effective way to increase the quit rate through using SC services.

Therefore, the present study will examine (1) the effectiveness of personalised active referral to smoking cessation (SC) services and text messaging on encouraging SC services (2) explore the use of CBPR model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

ELIGIBILITY:
Inclusion Criteria:

Hong Kong residents aged 18 or above

* Smoke at least 1 cigarette per day in the past 3 months
* Able to communicate in Cantonese
* Exhaled carbon monoxide (CO) 4 ppm or above, assessed by a validated CO smokerlyzer
* Have Intention to quit / reduce smoking

Exclusion Criteria:

* Smokers who have difficulties (either physical or cognitive condition) to communicate
* Currently following other smoking cessation programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
smoking quit rate change from baseline at 3-month follow-up | 3-month follow-up
  The primary outcomes are self-reported 7-day point prevalence (pp) quit rate at 3 month among the three groups
smoking quit rate change from baseline at 6-month follow-up | 6-month follow-up
  The primary outcomes are self-reported 7-day point prevalence (pp) quit rate at 3 month among the three groups

SECONDARY OUTCOMES:
Biochemical validated quit rate | 3-month follow-up
  biochemically validated quit rates at 3 month in the three groups
Biochemical validated quit rate | 6-month follow-up
  biochemically validated quit rates at 6 month in the three groups
Smoking reduction rate change from baseline at 3-month follow-up | 3-month follow-up
  rate of smoking reduction by at least half of baseline amount in the three groups
Smoking reduction rate change from baseline at 6-month follow-up | 6-month follow-up
  rate of smoking reduction by at least half of baseline amount in the three groups
Smoking quit attempt change from baseline at 3-month follow-up | 3-month follow-up
  number of quit attempts at 3 month among the three groups
Smoking quit attempt change from baseline at 6-month follow-up | 6-month follow-up
  number of quit attempts at 6 month among the three groups
quit rate for all subjects change from baseline at 3- and 6-month follow-up | 3 and 6 months follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2016
Reduction rate for all subjects change from baseline at 3- and 6-month follow-up | 3 and 6 months follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2016
Use of smoking cessation service | 3 and 6 months follow-up
  use of smoking cessation at 3 and 6 month follow-up among three groups
Use of smoking cessation service for all subjects | 3 and 6 months follow-up
  Use of smoking cessation service for all subjects participating in Quit to Win contest 2016

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Kelvin Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The Hong Kong Council on Smoking and Health (COSH), Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weng X, Wang MP, Suen YN, Li WHC, Wu Y, Cheung DYT, Kwong ACS, Lai VWY, Chan SSC, Lam TH. Comparing different intensities of active referral to smoking cessation services in promoting smoking cessation among community smokers: a study protocol of a cluster randomized controlled trial. BMC Public Health. 2018 Jul 4;18(1):830. doi: 10.1186/s12889-018-5782-1. PMID 29973191